CLINICAL TRIAL: NCT02962128
Title: Role of PUFA-Gene Interactions in Health Disparities
Brief Title: Role of Polyunsaturated Fatty Acids (PUFA)-Gene Interactions in Heath Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH); University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00038046; 1R01AT008621-01A1 (NIH)
Record Dates: First submitted 2016-10-25; First posted 2016-11-11 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2021-06

CONDITIONS: Fatty Acid-Gene Interactions
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Linoleic Acid (LA) Diet (Experimental): European Americans (genotypes: TT, GT & GG) and African Americans (genotypes: GT & GG) at rs173537will be randomly assigned to a high LA diet (10% energy) based on a randomized block design with 5 strata defined by race and genotype combinations.
  Interventions: Dietary Supplement: High Linoleic Acid (LA) Diet
- Low Linoleic Acid (LA) Diet (Experimental): European Americans (genotypes: TT, GT & GG) and African Americans (genotypes: GT & GG) at rs173537will be randomly assigned to a low LA diet (2.5% energy) based on a randomized block design with 5 strata defined by race and genotype combinations.
  Interventions: Dietary Supplement: Low Linoleic Acid (LA) Diet

INTERVENTIONS:
Dietary Supplement: High Linoleic Acid (LA) Diet — Volunteers will be randomly assigned to consumption of a high [10% energy] LA-containing diet for 12 weeks.
  Arms: High Linoleic Acid (LA) Diet
Dietary Supplement: Low Linoleic Acid (LA) Diet — Volunteers will be randomly assigned to consumption of a low [2.5% energy] LA-containing diet for 12 weeks.
  Arms: Low Linoleic Acid (LA) Diet

SUMMARY:
A randomized, clinical trial to provide the first comprehensive investigation of the role of fatty acid desaturate (FADS) genetic determinants on PUFA biosynthesis and metabolism as well as levels of inflammatory markers in a controlled dietary environment using two (low and high linoleic acid) parallel diets.

DETAILED DESCRIPTION:
Participants will be provided (weekly) with food items containing most of (>90%) the daily dietary fat (25-30% of daily calories) to be consumed. All study-supplied foods will be prepared by or acquired by the Wake Forest University Health Sciences (WFUHS) Clinical Research Unit (CRU) Metabolic Kitchen and distributed by the same. These foods will include smoothies (containing flaxseed oil common to both arms), and arm-dependent oil-based condiments (salad dressing, mayonnaise, and margarine) and prepared snack foods, each made with the arm-specific oil, as well as several packaged snacks and food items. Participants will be provided meal plans and recipes for home preparation of meals that will allow them to adhere to the target fatty acid contents of the two dietary arms. The goal of the dietary intervention is to provide participants with the daily fat content of their diet (25-30% of the daily calories) and to educate the participant to select and consume the balance of nutrients (60-75% of daily calories) derived from non-fat/low-fat containing foods.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Must agree to adhere to dietary intervention requirements during the entire 12-week study period
* Be willing to participate for the whole study
* Agree not to take any PUFA-based dietary supplements during the study
* Agree not to take interfering medications during the duration of the study
* Agree to allow samples to be stored for future use
* Self-identify as European American or African American

Exclusion Criteria:

* A diagnosis of diabetes, cancer, heart disease, arthrosclerosis, asthma, multiple sclerosis or chronic joint disease or the occurrence heart attack or vascular surgery within the past year, untreated high blood pressure or a history of stroke, having a pacemaker or a defibrillator
* use of tobacco products (smoked, smokeless, electronic) within the last six months
* Currently pregnant or lactating. Potential female subjects are asked in the telephone screening if they are pregnant or plan to become pregnant in the next year. Those answering in the affirmative are excluded. We will include in the Institutional Review Board (IRB) protocol and consent that subjects agree to use a reliable method of birth control during the time they are in the study.
* Having a current or recent history of eating disorders
* Having an allergy to safflower or, flaxseed or olive oils.
* fasting triglycerides (TG) greater than 150 mg/dl, as measured by Lab Corp at screening
* BP greater than 140/90 , as measured by a CRU nurse, at screening
* BMI equal to or greater than 30 or less than 19, as measured at screening
* fasting glucose greater than 125 mg/dl, as measured by Lab Corp at screening
* use of aspirin (>100 mg /day), NSAIDS or oral corticosteroids
* use of montelukast-type of allergy medications
* use of statins, niacin or fibrates or other lipid lowering medications
* use of botanical/fish (PUFA-containing) oil or dietary supplements for one month prior to joining the study .
* individuals not self-identifying as European American or African American
* individuals self-identifying as Hispanic
* Individuals of vulnerable populations, including children, will not be recruited for this study
* having an hsCRP measurement in excess of 3.0 at Visit 1

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Measurement in Change of PUFAs | 12 Weeks for Each Volunteer
  The primary outcome is the measurement of the change in PUFAs at 12 weeks. Biological specimens (urine and blood) will be collected from each subject at the beginning of the dietary intervention and at 4 week intervals. The primary outcome will be the measured difference between baseline and final PUFA levels before and after the diet.

SECONDARY OUTCOMES:
Measurement of Change in Serum Lipids (Cholesterol and Triglycerides) | 12 Weeks for Each Volunteer
  Secondary outcomes will be quantified in mg/dL and assessed using standard methods in an accredited clinical laboratory.

OTHER OUTCOMES:
Measurement of Change in Inflammatory Biomarkers (including Cytokines) | 12 Weeks for Each Volunteer
  The biochemical endpoints will be measured using established protocols

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sergeant, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen ST. Regulation of research: is it a drug trial or a supplement trial? Fitoterapia. 2011 Jan;82(1):14-6. doi: 10.1016/j.fitote.2010.11.011. Epub 2010 Nov 10. PMID 21073930
- [Background] Schaeffer L, Gohlke H, Muller M, Heid IM, Palmer LJ, Kompauer I, Demmelmair H, Illig T, Koletzko B, Heinrich J. Common genetic variants of the FADS1 FADS2 gene cluster and their reconstructed haplotypes are associated with the fatty acid composition in phospholipids. Hum Mol Genet. 2006 Jun 1;15(11):1745-56. doi: 10.1093/hmg/ddl117. Epub 2006 May 2. PMID 16670158
- [Background] Mathias RA, Sergeant S, Ruczinski I, Torgerson DG, Hugenschmidt CE, Kubala M, Vaidya D, Suktitipat B, Ziegler JT, Ivester P, Case D, Yanek LR, Freedman BI, Rudock ME, Barnes KC, Langefeld CD, Becker LC, Bowden DW, Becker DM, Chilton FH. The impact of FADS genetic variants on omega6 polyunsaturated fatty acid metabolism in African Americans. BMC Genet. 2011 May 20;12:50. doi: 10.1186/1471-2156-12-50. PMID 21599946
- [Background] Sergeant S, Hugenschmidt CE, Rudock ME, Ziegler JT, Ivester P, Ainsworth HC, Vaidya D, Case LD, Langefeld CD, Freedman BI, Bowden DW, Mathias RA, Chilton FH. Differences in arachidonic acid levels and fatty acid desaturase (FADS) gene variants in African Americans and European Americans with diabetes or the metabolic syndrome. Br J Nutr. 2012 Feb;107(4):547-55. doi: 10.1017/S0007114511003230. Epub 2011 Jul 4. PMID 21733300
- [Background] Malerba G, Schaeffer L, Xumerle L, Klopp N, Trabetti E, Biscuola M, Cavallari U, Galavotti R, Martinelli N, Guarini P, Girelli D, Olivieri O, Corrocher R, Heinrich J, Pignatti PF, Illig T. SNPs of the FADS gene cluster are associated with polyunsaturated fatty acids in a cohort of patients with cardiovascular disease. Lipids. 2008 Apr;43(4):289-99. doi: 10.1007/s11745-008-3158-5. Epub 2008 Mar 5. PMID 18320251
- [Background] Xie L, Innis SM. Genetic variants of the FADS1 FADS2 gene cluster are associated with altered (n-6) and (n-3) essential fatty acids in plasma and erythrocyte phospholipids in women during pregnancy and in breast milk during lactation. J Nutr. 2008 Nov;138(11):2222-8. doi: 10.3945/jn.108.096156. PMID 18936223
- [Background] Lattka E, Koletzko B, Zeilinger S, Hibbeln JR, Klopp N, Ring SM, Steer CD. Umbilical cord PUFA are determined by maternal and child fatty acid desaturase (FADS) genetic variants in the Avon Longitudinal Study of Parents and Children (ALSPAC). Br J Nutr. 2013 Apr 14;109(7):1196-210. doi: 10.1017/S0007114512003108. Epub 2012 Aug 9. PMID 22877655
- [Background] Bokor S, Dumont J, Spinneker A, Gonzalez-Gross M, Nova E, Widhalm K, Moschonis G, Stehle P, Amouyel P, De Henauw S, Molnar D, Moreno LA, Meirhaeghe A, Dallongeville J; HELENA Study Group. Single nucleotide polymorphisms in the FADS gene cluster are associated with delta-5 and delta-6 desaturase activities estimated by serum fatty acid ratios. J Lipid Res. 2010 Aug;51(8):2325-33. doi: 10.1194/jlr.M006205. Epub 2010 Apr 28. PMID 20427696
- [Background] Ramsden CE, Zamora D, Leelarthaepin B, Majchrzak-Hong SF, Faurot KR, Suchindran CM, Ringel A, Davis JM, Hibbeln JR. Use of dietary linoleic acid for secondary prevention of coronary heart disease and death: evaluation of recovered data from the Sydney Diet Heart Study and updated meta-analysis. BMJ. 2013 Feb 4;346:e8707. doi: 10.1136/bmj.e8707. PMID 23386268
- [Background] Chilton FH, Murphy RC, Wilson BA, Sergeant S, Ainsworth H, Seeds MC, Mathias RA. Diet-gene interactions and PUFA metabolism: a potential contributor to health disparities and human diseases. Nutrients. 2014 May 21;6(5):1993-2022. doi: 10.3390/nu6051993. PMID 24853887
- [Background] Mathias RA, Pani V, Chilton FH. Genetic Variants in the FADS Gene: Implications for Dietary Recommendations for Fatty Acid Intake. Curr Nutr Rep. 2014 Jun;3(2):139-148. doi: 10.1007/s13668-014-0079-1. PMID 24977108
- [Background] Ramsden CE, Faurot KR, Zamora D, Suchindran CM, MacIntosh BA, Gaylord S, Ringel A, Hibbeln JR, Feldstein AE, Mori TA, Barden A, Lynch C, Coble R, Mas E, Palsson O, Barrow DA, Mann DJ. Targeted alteration of dietary n-3 and n-6 fatty acids for the treatment of chronic headaches: a randomized trial. Pain. 2013 Nov;154(11):2441-2451. doi: 10.1016/j.pain.2013.07.028. Epub 2013 Jul 22. PMID 23886520

DOCUMENTS (1):
  • Informed Consent Form (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT02962128/ICF_000.pdf